CLINICAL TRIAL: NCT02273635
Title: Controlled, Randomized, Double-blind Clinical Trial, 24 Months Duration, to Compare the Efficacy, Safety and Tolerability of Andrographolide Versus Placebo in Patients With Progressive Forms of Multiple Sclerosis
Brief Title: Efficacy, Safety and Tolerability of Andrographolides Versus Placebo in Patients With Progressive Forms of MS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innobioscience SpA (Industry)
Collaborators: Pontificia Universidad Catolica de Chile (Other); University of Chile (Other); Universidad Austral de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14PIE-26946CORFO; 14-391 (Other: Comite Etico Cientifico - CEC MED UC)
Record Dates: First submitted 2014-10-03; First posted 2014-10-24 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Primary Progressive Multiple Sclerosis; Multiple Sclerosis, Secondary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — andrographolide; neoandrographolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- andrographolides (Experimental): Coated tablets containing 140 mg andrographolides twice a day orally administered for a period of 24 months.
  Interventions: Drug: Andrographolides
- sugar tablets (Placebo Comparator): Coated tablets containing 140 mgs excipients twice a day orally administered for a period of 24 months.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Andrographolides — 140 mg andrographolides coated tablets twice a day orally administered for 24 months.
  Other Names: andrographolide, neoandrographolide, deoxyandrographolide; IB-MS 14
  Arms: andrographolides
Drug: placebo — 140 mg excipients coated tablets twice a day orally administered for 24 months
  Arms: sugar tablets

SUMMARY:
The purpose of this study is to compare the efficacy and safety of andrographolide 140 mg administered twice a day orally versus a placebo as a modifying treatment of the disease in patients with the progressive forms of Multiple Sclerosis (MS).

The principal outcome is to determine the efficacy, of andrographolide in retarding the progression of brain atrophy in patients with progressive forms of MS.

DETAILED DESCRIPTION:
1. Evaluate the clinical efficacy of andrographolide 140 mg administered orally twice a day versus a placebo in:

   * Delay in the disability capacity progression through the Expanded Disability Status Scale (EDSS) and Multiple Sclerosis Functional Composite (MSFC) at 24 months compared to the baseline.
   * Delay in cognitive impairment by means of Paced Auditory Serial Addition Test (PASAT), Symbol Digit Modalities Test (SDMT) and depression (Beck) at 24 months compared to the baseline.
   * Quality of life Multiple Sclerosis Impact Scale (MSIS 29) and fatigue (Krupp) through parameters reported by the patients at at 24 months compared to the baseline.
   * Tolerability of andrographolide measured by the Treatment Satisfaction Questionnaire for Medication (TSQM) at 24 months.
   * Delay in the decrease in brain volume measured by Magnetic Resonance (MR) at 24 months compared to the baseline.
   * Number and volume of new lesions or larger size in T2 by MR at 24 months compared to the baseline.
   * Number of new hipointense lesions in T1 or (gadolinium captive) by MR at 24 months compared to the baseline.
   * Delay in the retineal thinning measured by Optical Coherence Tomography (OCT) and visual field at 24 months compared to the baseline.
   * Safety of andrographolide at 24 months through the record of adverse effects in symptom dairy and programmed interviews.
2. Explore the pharmacokinetic of andrographolide 140 mg administered orally twice day in:

   * bio availability and concentration of andrographolide in the patients with treatment.
   * half-life, maximum concentration, clearance of andrographolide in equilibrium state.
3. Determine the immunomodulatory effects of andrographolide 140 mg administered twice a day orally on lymphocyte populations in patients through the:

   * Determination of Th1, Th2, Th17 and Treg lymphocyte sub-populations.
   * Determination of cytokines IFNgama, TNFalpha, IL2, IL17alpha and TGFbeta.

Population: adult patients, men and women with progressive forms of MS. The number of patients to be selected will be 68, to randomly assign 34 patients to each group.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent previous to the initiation of the study before any evaluation.
* Men and women > 18 years of age with Minimental > 24.
* Patients with diagnosis of secondary progressive MS without relapses or primary progressive MS according to the criteria of McDonald 2010.

Exclusion Criteria:

* Relapsing-remitting MS
* Current Immunomodulatory or immunosuppressive therapy
* Uncontrolled systemic diseases not controlled or treated with immunotherapy (i.e Rheumatoid Arthritis, Lupus Erythematosus).
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-11 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Brain atrophy in patients with progressive forms of MS | 24 months
  Retarding the progression of brain atrophy as measured by MR quantified by the percentage of change in volume size utilizing SIENA.

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | 24 months
  Delay in the disability capacity progression through the Expanded Disability Status Scale (EDSS) at 24 months compared to the baseline.
Paced Auditory Serial Addition Test (PASAT) | 24 months
  Delay in cognitive impairment by means of Paced Auditory Serial Addition Test (PASAT) at 24 months compared to the baseline.
Quality of life Multiple Sclerosis Impact Scale (MSIS 29) | 24 months
  Quality of life Multiple Sclerosis Impact Scale (MSIS 29) through parameters reported by the patients at 24 months compared to the baseline.
Treatment Satisfaction Questionnaire for Medication (TSQM) | 24 months
  Tolerability of andrographolide measured by the Treatment Satisfaction Questionnaire for Medication (TSQM) at 24 months.
Number of new T2 lesions | 24 months
  Number of new lesions T2 by MR at 24 months compared to the baseline.
New hypointense lesions in T1 | 24 months
  Number of new hypointense lesions in T1 by MR at 24 months compared to the baseline.
Optical Coherence Tomography (OCT) | 24 months
  Delay in the retinal thinning measured by Optical Coherence Tomography (OCT) at 24 months compared to the baseline.
Record of adverse effects in daily symptoms and programmed interviews. | 24 months
  Safety of andrographolide at 24 months through the record of adverse effects in daily symptoms and programmed interviews.
Multiple Sclerosis Functional Composite (MSFC) | 24 months
  Delay in the disability capacity progression through the Multiple Sclerosis Functional Composite (MSFC) at 24 months compared to the baseline.
Symbol Digit Modalities Test (SDMT) | 24 months
  Delay in cognitive impairment by means of Symbol Digit Modalities Test (SDMT) at 24 months compared to the baseline.
Depression by Beck scale | 24 months
  Evaluate mood disorders by means of Beck scale at 24 months compared to the baseline.
Fatigue by Krupp scale | 24 months
  Evaluate fatigue by Krupp scale reported by the patients at 24 months compared to the baseline.
Number of new gadolinium enhancement lesions in T1 by MR | 24 months
  Number of new gadolinium enhancement lesions in T1 by MR at 24 months compared to the baseline.
Visual field | 24 months
  Change in visual field at 24 months compared to the baseline.
Volume of new T2 lesions | 24 months
  Volume of size in T2 by MR at 24 months compared to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Juan L Hancke, DVM, PhD, Study Director — Universidad Austral de Chile
Locations (1):
- Multiple Sclerosis Centre, Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Iruretagoyena MI, Tobar JA, Gonzalez PA, Sepulveda SE, Figueroa CA, Burgos RA, Hancke JL, Kalergis AM. Andrographolide interferes with T cell activation and reduces experimental autoimmune encephalomyelitis in the mouse. J Pharmacol Exp Ther. 2005 Jan;312(1):366-72. doi: 10.1124/jpet.104.072512. Epub 2004 Aug 26. PMID 15331658
- [Background] Iruretagoyena MI, Sepulveda SE, Lezana JP, Hermoso M, Bronfman M, Gutierrez MA, Jacobelli SH, Kalergis AM. Inhibition of nuclear factor-kappa B enhances the capacity of immature dendritic cells to induce antigen-specific tolerance in experimental autoimmune encephalomyelitis. J Pharmacol Exp Ther. 2006 Jul;318(1):59-67. doi: 10.1124/jpet.106.103259. Epub 2006 Apr 5. PMID 16597709
- [Background] Burgos RA, Hancke JL, Bertoglio JC, Aguirre V, Arriagada S, Calvo M, Caceres DD. Efficacy of an Andrographis paniculata composition for the relief of rheumatoid arthritis symptoms: a prospective randomized placebo-controlled trial. Clin Rheumatol. 2009 Aug;28(8):931-46. doi: 10.1007/s10067-009-1180-5. Epub 2009 Apr 29. PMID 19408036
- [Background] Cabrera D, Gutierrez J, Cabello-Verrugio C, Morales MG, Mezzano S, Fadic R, Casar JC, Hancke JL, Brandan E. Andrographolide attenuates skeletal muscle dystrophy in mdx mice and increases efficiency of cell therapy by reducing fibrosis. Skelet Muscle. 2014 Mar 21;4:6. doi: 10.1186/2044-5040-4-6. eCollection 2014. PMID 24655808
- [Background] Carretta MD, Alarcon P, Jara E, Solis L, Hancke JL, Concha II, Hidalgo MA, Burgos RA. Andrographolide reduces IL-2 production in T-cells by interfering with NFAT and MAPK activation. Eur J Pharmacol. 2009 Jan 14;602(2-3):413-21. doi: 10.1016/j.ejphar.2008.11.011. Epub 2008 Nov 13. PMID 19038244
- [Background] Burgos RA, Seguel K, Perez M, Meneses A, Ortega M, Guarda MI, Loaiza A, Hancke JL. Andrographolide inhibits IFN-gamma and IL-2 cytokine production and protects against cell apoptosis. Planta Med. 2005 May;71(5):429-34. doi: 10.1055/s-2005-864138. PMID 15931581
- [Background] Hidalgo MA, Romero A, Figueroa J, Cortes P, Concha II, Hancke JL, Burgos RA. Andrographolide interferes with binding of nuclear factor-kappaB to DNA in HL-60-derived neutrophilic cells. Br J Pharmacol. 2005 Mar;144(5):680-6. doi: 10.1038/sj.bjp.0706105. PMID 15678086
- [Background] Sandborn WJ, Targan SR, Byers VS, Rutty DA, Mu H, Zhang X, Tang T. Andrographis paniculata extract (HMPL-004) for active ulcerative colitis. Am J Gastroenterol. 2013 Jan;108(1):90-8. doi: 10.1038/ajg.2012.340. Epub 2012 Oct 9. PMID 23044768
- [Background] Tang T, Targan SR, Li ZS, Xu C, Byers VS, Sandborn WJ. Randomised clinical trial: herbal extract HMPL-004 in active ulcerative colitis - a double-blind comparison with sustained release mesalazine. Aliment Pharmacol Ther. 2011 Jan;33(2):194-202. doi: 10.1111/j.1365-2036.2010.04515.x. Epub 2010 Nov 30. PMID 21114791
- [Derived] Ciampi E, Uribe-San-Martin R, Carcamo C, Cruz JP, Reyes A, Reyes D, Pinto C, Vasquez M, Burgos RA, Hancke J. Efficacy of andrographolide in not active progressive multiple sclerosis: a prospective exploratory double-blind, parallel-group, randomized, placebo-controlled trial. BMC Neurol. 2020 May 7;20(1):173. doi: 10.1186/s12883-020-01745-w. PMID 32380977